CLINICAL TRIAL: NCT01961557
Title: Evaluating an Extension Assist Knee Ankle Foot Orthosis to Improve Gait in Children With Movement Disorders
Brief Title: Evaluating a New Knee-Ankle-Foot Brace to Improve Gait in Children With Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 130210; 13-CC-0210
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-07-17

CONDITIONS: Incomplete Spinal Cord Injury; Muscular Dystrophy; Spina Bifida; Cerebral Palsy
Keywords: incomplete spinal cord injury; EEG; Cerebral Palsy; Knee; Muscular Dystrophies
MeSH Terms: conditions — Muscular Dystrophies; Spinal Dysraphism; Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- There is a single study arm in this feasibility study. (Experimental): All participants will be evaluated using the different configurations of the EA-KAFO (see Table 1 in the protocol), which includes the configuration that contains the Active Motorized KAFO and the configuration that contains the Powerwalk Knee Exoskeleton. Each subject will serve as their own control to assess the effect of each configuration of the EA-KAFO interventions.
  Interventions: Device: EA-KAFO

INTERVENTIONS:
Device: EA-KAFO — This study tests a single device that contains multiple potential configurations as outlined in Table 1 of the protocol. Each participant be evaluated in multiple configurations, minimally including the baseline configuration and the motor assist condition at the knee.

SUMMARY:
Background:

- Cerebral palsy (CP) is the most common motor disorder in children. CP often causes crouch gait, an abnormal way of walking. Knee crouch has many causes, so no single device or approach works best for everybody. This study s adjustable brace provides many types of walking assistance. Researchers will evaluate brace options to find the best solution for each participant, and whether one solution works best for the group.

Objective:

- To evaluate a new brace to improve crouch gait in children with CP.

Eligibility:

* Children 5 17 years old with CP.
* Healthy volunteers 5 17 years old.

Design:

* All participants will be screened with medical history and physical exam.
* Healthy volunteers will have 1 visit. They will do motion analysis, EMG, and EEG described below.
* Participants with CP will have 6 visits.
* Visit 1:

<TAB>1. Motion analysis: Balls will be taped to participants skin. This helps cameras follow their movement.

<TAB>2. EMG: Metal discs will be taped to participants skin. They measure electrical muscle activity.

<TAB>3. Participants knee movement will be tested.

<TAB>4. Participants will walk 50 meters.

<TAB>5. Participants legs will be cast to make custom braces.

* Visit 2:
* Participants will wear their new braces and have them adjusted.
* Steps 1 3 will be repeated.
* EEG: Small metal discs will be placed on the participants scalp. They record brain waves.
* Participants will have electrical stimulation of their knees and practice extending them.
* Participants will take several walks with the braces in different settings.
* Visits 3 5: participants will repeat the walking and some other steps from visit 2.
* Visit 6 will repeat visit 2.

DETAILED DESCRIPTION:
Objective

The purpose of this protocol is to evaluate several configurations of a prototype Extension Assist Knee-Ankle-Foot Orthosis (EA-KAFO) in patients with cerebral palsy (CP), muscular dystrophy (MD), spina bifida (SB), or incomplete spinal cord injury (iSCI) who have knee extension deficiency. Three forms of assistance will be provided at the knee joint including a passive-damper component, functional electrical stimulation (FES) to the quadriceps, and a motorized assist. One form will provide controllable resistance at the knee to strengthen muscles and promote knee extension after the resistance is removed. These will be compared to traditional bracing which typically improves crouch by blocking some or all motion at one or both joints. We hypothesize that all assistive configurations will improve gait alignment and performance compared to the non-assisted conditions. We further hypothesize that a best solution for each participant will exist, but may vary across subjects due to the heterogeneity of these movement disorders. Preliminary data on brain activation using EEG will be collected during all walking conditions.

Study population

Thirty (30) subjects, age 5 and above, diagnosed with crouch gait from diplegic CP, (30) subjects, age 5 and above, with knee extension deficiency from MD, SB, or iSCI (15 from each group) and 10 age-matched healthy volunteers will be recruited.

Design

This protocol will evaluate an EA-KAFO prototype consisting of a custom fabricated brace combined with a modular knee joint with three modes of operation: hinge (no assist), a passive spring-damper, and an active motorized assist. Since crouch can also be precipitated at the ankle, the orthotic ankle joint has an adjustable dynamic resistance (ADR) mechanism that can be locked (passive assist) to simulate a standard brace, free, or provide variable resistance to assist knee extension. Additionally, we will combine quadriceps FES with the hinge and the passive damper to create two hybrid configurations. The hinge and the passive damper (Ultraflex ) knee modules, and ADR ankle brace are FDA-approved (Class I), commercially available devices. This protocol for evaluation of the active motorized joint module, the two hybrid configurations, and the controllable resistance device (PowerWalk by Agilik Technologies) has been reviewed by the FDA as a medical device study and was determined by the FDA to be non-significant risk. Healthy controls will come for one visit, and participants with movement disorders will complete 6-10 visits: 1) initial assessment and casting for custom leg brace; 2) EA-KAFO configuration; 3) initial data collection and practice; 4-5) accommodation to brace configurations; 6) final data collection. Additional accommodation visits may be added if necessary, up to the maximum of 10 total visits. Participants with movement disorders will be permitted to re-enroll in the protocol is a minimum of 1 year has passed from their prior final visit. Motion capture, force plates, and electromyography (EMG) will be used for gait analysis while electroencephalography (EEG) will measure brain activity during walking.

Outcome measures

The primary outcome is the amount of knee flexion during gait. The optimal solution for each individual will be that which provides the greatest reduction in peak knee angle. Secondary outcomes will include gait speed, knee extensor moment, and EEG activation profiles.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 5 years and above
* Either a healthy volunteer, have crouch gait with a diagnosis of spastic diplegic cerebral palsy, or have lower extremity weakness resulting in gait pathology from a diagnosis of muscular dystrophy, spina bifida, or incomplete spinal cord injury.
* Able to understand and follow simple directions based on parent report and physician observation during history and physical examination.
* Able to provide verbal/written assent.
* Less than 5 degrees of knee flexion contracture with hip extended in supine position. Hamstring contracture as assessed by straight leg raising test does not limit ability to participate in the study.
* Less than 10 degrees of plantar flexion contracture in neutral foot alignment.
* A measured foot-thigh angle of -10 to 25 degrees in prone position.
* Diagnosed with knee extension deficiency as indicated by a crouched posture during gait lacking at least 20 degrees of knee extension at mid stance during walking as assessed visually, knee extensor muscle weakness which prevents full extension of the limb, or reliance upon braces or other aids which lock the knee during walking. (The exact level of knee extension deficiency, or crouch, will be quantified after inclusion using gait analysis.)
* Able to walk at least 10 feet without stopping with or without a walking aid
* Agreement to not drink caffeine for 24 hours before each EEG assessment (CP only) visit because it can modify brain activity

EXCLUSION CRITERIA:

* Any neurological, musculoskeletal or cardiorespiratory injury, health condition, or diagnosis other than cerebral palsy, muscular dystrophy, spina bifida, or incomplete spinal cord injury that would affect the ability to walk as directed for short periods of time.
* Participation in this protocol within the previous 1 year.

ADDITIONAL EXCLUSION CRITERIA FOR INDIVIDUALS WITH CEREBRAL PALSY:

* A history of a seizure in the past year.
* Pregnancy

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Peak knee angle | This outcome will be assessed twice, at the initial and final data assessment visits, as indicated in the protocol.
  The primary outcome measure will be the effect of the intervention on crouch, as measured by peak knee angle during walking with the EA-KAFO. the outcome description refers to the general Extension Assist Knee Ankle Foot Orthosis (EA-KAFO). The outcome measure will be assessed across the different configurations of the EA-KAFO, which includes the configuration that contains the Active Motorized KAFO and the configuration that contains the Powerwalk Knee Exoskeleton.

SECONDARY OUTCOMES:
Secondary outcome measures | At the same time
  Secondary outcome measures, assessed at the same time frame and across the same configurations of the EA-KAFO as the primary outcome measure, include Gait Speed and Knee Joint Moment.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Bulea, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent about sharing IPD.

REFERENCES:
- [Background] Molnar GE. Rehabilitation in cerebral palsy. West J Med. 1991 May;154(5):569-72. PMID 1866952
- [Background] Yeargin-Allsopp M, Van Naarden Braun K, Doernberg NS, Benedict RE, Kirby RS, Durkin MS. Prevalence of cerebral palsy in 8-year-old children in three areas of the United States in 2002: a multisite collaboration. Pediatrics. 2008 Mar;121(3):547-54. doi: 10.1542/peds.2007-1270. PMID 18310204
- [Background] Binder H, Eng GD. Rehabilitation management of children with spastic diplegic cerebral palsy. Arch Phys Med Rehabil. 1989 Jun;70(6):482-9. doi: 10.1016/0003-9993(89)90012-9. PMID 2658915
- [Derived] Shideler BL, Bulea TC, Chen J, Stanley CJ, Gravunder AJ, Damiano DL. Toward a hybrid exoskeleton for crouch gait in children with cerebral palsy: neuromuscular electrical stimulation for improved knee extension. J Neuroeng Rehabil. 2020 Sep 3;17(1):121. doi: 10.1186/s12984-020-00738-7. PMID 32883297
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-CC-0210.html